CLINICAL TRIAL: NCT00142337
Title: A Phase 2, One Arm, Open Label, Feasibility Study Assessing One Month Zidovudine/Didanosine Postpartum Prophylaxis to Prevent Resistance Mutations in Mothers Exposed to Single Dose Nevirapine to Prevent Mother to Child Transmission of HIV
Brief Title: One Month Dual Antiretroviral Prophylaxis to Prevent Resistance Mutations in Mothers Exposed to Single Dose Nevirapine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Responsible Party: Principal Investigator, Marc Lallemant, Senior Researcher, Institut de Recherche pour le Developpement
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IRD-UMI 174 PHPT-4
Record Dates: First submitted 2005-09-01; First posted 2005-09-02 (Estimated); Last update posted 2012-01-06 (Estimated); Status verified 2012-01

CONDITIONS: HIV Infections
Keywords: zidovudine; didanosine; Prevention of mother to child transmission of HIV; nevirapine; Thailand; Resistance; HIV; Postpartum period
MeSH Terms: conditions — HIV Infections | interventions — Zidovudine; Didanosine

INTERVENTIONS:
Drug: Zidovudine (ZDV) — Zidovudine 300 mg, twice daily, for one month postpartum. Note: after July 03, 2005, all women received 200 mg, twice daily, for the same duration.
Drug: Didanosine (ddI) — 250 mg ddI-EC (400 mg if body weight >60 kg) once daily, starting at the onset of labor and for one month postpartum

SUMMARY:
The purpose of this study is to determine whether providing zidovudine (ZDV) and didanosine (ddI) during labor and for one month postpartum can reduce the selection of nevirapine (NVP) resistance mutations postpartum in women who received a single dose of nevirapine during labor and standard ZDV prophylaxis for the prevention of mother to child transmission of HIV.

DETAILED DESCRIPTION:
A single nevirapine dose to the mother, with or without a dose to the child, in addition to oral ZDV prophylaxis starting from 28 weeks gestation has been proven to be highly effective in reducing further mother-to-child HIV transmission (PMTCT).

However, post exposure nevirapine resistance mutations are observed in the mother's viral population. These mutations detectable very early after exposure tend to disappear over time.

Nevertheless, they may be associated with decrease in efficacy of non-nucleoside reverse transcriptase inhibitor (NNRTI) containing regimens subsequently given to the women for their own health.

Therefore, there is a need for research to prevent selection of resistance in the first place or to overcome the resistance in subsequent treatment of the infected mother or infant.

Nevirapine plasma levels above IC50 have been detected in women exposed to a single 200 mg dose of nevirapine in a significant number of women during the third week postpartum.

We hypothesize that giving ZDV+ddI to women exposed to nevirapine for one month as soon as possible after exposure may prevent the selection of nevirapine resistance mutations.

ELIGIBILITY:
Inclusion Criteria:

* Meet all pre-entry criteria;
* Consent to participate and to be followed for the duration of the study;
* Present the following laboratory values within 14 days prior to inclusion:

  * Hemoglobin > 8.0 mg/dl
  * Absolute neutrophil count > 1000 cells/mm3
  * Platelets > 100,000 cells/mm3
  * Serum creatinine < 1.5 mg/dl (women with a serum creatinine > 1.5 mg/dl must have a measured eight-hour urine creatinine clearance > 70 ml/min)
  * SGPT less than 10 times the upper limit of normal
  * Amylase less than 150/L IU (this upper limit may change slightly depending on the normal range at the hospital laboratory).

Exclusion Criteria:

* Evidence of pre-existing fetal anomalies incompatible with life;
* Known hypersensitivity to any benzodiazepine or to NVP;
* Receipt of antiretroviral agent other than ZDV;
* Receipt of non-allowed concomitant treatment or contraindication to ddI
* Concurrent participation in another clinical trial;
* Women with a CD4 count <200/µL or history of oral candidiasis if they are not receiving pneumocystis carinii pneumonia (PCP) prophylaxis
* Any other contra-indicated drugs during ZDV+ddI treatment for the mother as well as the child (Contra-indicated drugs such as gancyclovir, isoniazid, linezolid, ethambutol, rifabutin, cidofovir are not allowed during the ZDV ddI treatment after delivery in order to prevent pharmacological interactions or overlapping toxicities.)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2004-12; Primary Completion 2006-05 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with viral NNRTI mutations detectable during the 4 month follow-up compared with the incidence observed in the PHPT-2 clinical trial, who received the same antiretroviral prophylaxis but no post-partum regimen | Within 4 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Marc Lallemant, MD, Principal Investigator — Institut de Recherche pour le Developpement
Locations (32):
- Thailand (32):
  - Bhumibol Adulyadej Hospital, Bangkok, Bangkok
  - Health Promotion Hospital Regional Center I, Bangkok, Bangkok
  - Chacheongsao Hospital, Muang, Chacheongsao
  - Prapokklao Hospital, Muang, Changwat Chanthaburi
  - Mae Chan Hospital, Mae Chan, Changwat Chiang Rai
  - Mae Sai Hospital, Mae Sai, Changwat Chiang Rai
  - Phan Hospital, Phan, Changwat Chiang Rai
  - Somdej Pranangchao Sirikit Hospital, Chon Buri, Changwat Chon Buri
  - Chonburi Hospital, Muang, Changwat Chon Buri
  - Kalasin Hospital, Muang, Changwat Kalasin
  - Kranuan Crown Prince Hospital, Kranuan, Changwat Khon Kaen
  - Khon Kaen Hospital, Muang, Changwat Khon Kaen
  - Regional Health Promotion Centre 6, Khon Kaen, Muang, Changwat Khon Kaen
  - Srinagarind Hospital, Muang, Changwat Khon Kaen
  - Lampang Hospital, Muang, Changwat Lampang
  - Nong Khai Hospital, Muang, Changwat Nong Khai
  - Pranangklao Hospital, Muang, Changwat Nonthaburi
  - Chiang Kham Hospital, Chiang Kham, Changwat Phayao
  - Buddhachinaraj Hospital, Muang, Changwat Phitsanulok
  - Ratchaburi Hospital, Muang, Changwat Ratchaburi
  - Rayong Hospital, Muang, Changwat Rayong
  - Roi-et Hospital, Muang, Changwat Roi Et
  - Hat Yai Hospital, Hat Yai, Changwat Songkhla
  - Nakornping Hospital, Mae Rim, Chiang Mai
  - Health Promotion Center Region 10, Muang, Chiang Mai
  - Lamphun Hospital, Munag, Chiang Mai
  - Chiangrai Prachanukroh Hospital, Muang, Chiangrai
  - Phaholpolphayuhasena Hospital, Munag, Kanchanaburi
  - Nakhonpathom Hospital, Muang, Nakhonpathom
  - Maharaj Nakornratchasrima Hospital, Muang, Nakornratchasrima
  - Samutprakarn Hospital, Samutprakarn, Samutprakarn
  - Samutsakorn Hospital, Muang, Samutsakorn

REFERENCES:
- [Background] Lallemant M, Jourdain G, Le Coeur S, Mary JY, Ngo-Giang-Huong N, Koetsawang S, Kanshana S, McIntosh K, Thaineua V; Perinatal HIV Prevention Trial (Thailand) Investigators. Single-dose perinatal nevirapine plus standard zidovudine to prevent mother-to-child transmission of HIV-1 in Thailand. N Engl J Med. 2004 Jul 15;351(3):217-28. doi: 10.1056/NEJMoa033500. Epub 2004 Jul 9. PMID 15247338
- [Background] Jourdain G, Ngo-Giang-Huong N, Le Coeur S, Bowonwatanuwong C, Kantipong P, Leechanachai P, Ariyadej S, Leenasirimakul P, Hammer S, Lallemant M; Perinatal HIV Prevention Trial Group. Intrapartum exposure to nevirapine and subsequent maternal responses to nevirapine-based antiretroviral therapy. N Engl J Med. 2004 Jul 15;351(3):229-40. doi: 10.1056/NEJMoa041305. Epub 2004 Jul 9. PMID 15247339
- [Background] Cressey TR, Jourdain G, Lallemant MJ, Kunkeaw S, Jackson JB, Musoke P, Capparelli E, Mirochnick M. Persistence of nevirapine exposure during the postpartum period after intrapartum single-dose nevirapine in addition to zidovudine prophylaxis for the prevention of mother-to-child transmission of HIV-1. J Acquir Immune Defic Syndr. 2005 Mar 1;38(3):283-8. PMID 15735445
- [Result] Lallemant M, Ngo-Giang-Huong N, Jourdain G, Traisaithit P, Cressey TR, Collins IJ, Jarupanich T, Sukhumanant T, Achalapong J, Sabsanong P, Chotivanich N, Winiyakul N, Ariyadej S, Kanjanasing A, Ratanakosol J, Hemvuttiphan J, Kengsakul K, Wannapira W, Sittipiyasakul V, Pornkitprasarn W, Liampongsabuddhi P, McIntosh K, Van Dyke RB, Frenkel LM, Koetsawang S, Le Coeur S, Kanchana S; PHPT-4 Study Team. Efficacy and safety of 1-month postpartum zidovudine-didanosine to prevent HIV-resistance mutations after intrapartum single-dose nevirapine. Clin Infect Dis. 2010 Mar 15;50(6):898-908. doi: 10.1086/650745. PMID 20158398